CLINICAL TRIAL: NCT02131207
Title: Novel Screening MRI for the Detection of Prostate Cancer
Brief Title: MRI Before Biopsy in Diagnosing Patients With Prostate Cancer
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator Left Institution
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE6813; NCI-2014-00822 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE6813 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-04-17; First posted 2014-05-06 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Diagnostic (MRI and biopsy): Participants undergo pelvic magnetic resonance imaging (MRI). Within 1-2 weeks, patients undergo scheduled prostate biopsy.
  Interventions: Device: magnetic resonance imaging; Procedure: prostate biopsy

INTERVENTIONS:
Device: magnetic resonance imaging — Undergo pelvic MRI
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
Procedure: prostate biopsy — Undergo prostate biopsy
  Other Names: biopsy of prostate; prostatic biopsy

SUMMARY:
This pilot clinical trial studies how well magnetic resonance imaging (MRI) before biopsy works in diagnosing patients with prostate cancer. MRI is a procedure in which radio waves and a powerful magnet linked to a computer are used to create detailed pictures of areas inside the body. This diagnostic procedure may aid in identifying lesions in the prostate which may have cancer. The lesions can then be targeted during the prostate biopsy to improve the accuracy of identifying prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identification of one of more lesions suspicious for prostate cancer using a novel MRI protocol, not identified by transrectal ultrasound (TRUS) alone and to determine if the lesions identified by MRI demonstrate clinically significant prostate cancer based on pathologic findings (ie. Gleason >= 7 or percentage of core involved with cancer > 50%).

SECONDARY OBJECTIVES:

I. Average time for MRI scan per patient. II. Correlation of lesions on MRI to radical prostatectomy specimens. III. To determine whether MRI 3 dimensional (3D) T2 half-Fourier acquired single turbo spin-echo (HASTE) or sampling perfection with application optimized contrast using different flip angle evolutions (SPACE) protocols provide improved rates of prostate cancer detection.

IV. Yield of additional clinically significant prostate cancer diagnoses based on MRI targeted lesions on biopsy.

V. Rate of benign pathology identified by MRI (i.e. false positives). VI. To compare costs associated with the use of MRI over TRUS biopsy alone.

OUTLINE:

Participants undergo pelvic MRI. Within 1-2 weeks, patients undergo scheduled prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal prostate-specific antigen (PSA) blood test

  * > 2.5 ng/mL for men < 50 years (yrs) of age
  * > 3.5 ng/mL for men < 60 yrs of age
  * > 4.5 ng/mL for men < 70 yrs of age
* Abnormal digital rectal exam (i.e. palpable nodule, induration or firm area to the prostate)
* Scheduled for a TRUS biopsy based on clinical suspicion for prostate cancer

Exclusion Criteria:

* Individuals who have previously undergone biopsy of the prostate for diagnosis of prostate cancer
* Contraindications to TRUS/prostate biopsy (BX)

  * Currently on blood thinning agents (Plavix, Coumadin etc.) or bleeding disorder
  * Active urinary tract infection
  * Acute painful perianal disorder (i.e. rectal abscess)
* Contraindications to MRI

  * Patients with ferromagnetic or otherwise non-MRI compatible aneurysm clips
  * The presence of an implanted pacemaker or implanted defibrillator device
  * Patients with contraindications for MRI due to embedded foreign metallic objects: bullets, shrapnel, metalwork fragments, or other metallic material adds unnecessary risk to the patient
  * Implanted medical device not described above that is not MRI-compatible
  * Known history of claustrophobia
* Individuals with a short life expectancy (< 10 years)

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a pilot study of patients from the University Hospitals urology clinics who have not previously been given a diagnosis of prostate cancer but who are awaiting a prostate biopsy due to an elevated PSA or abnormal digital rectal exam
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2014-09-10 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Increased detection of clinically significant prostate cancer | Up to 1 year
  Percent increase of patients with positive prostate cancer biopsies detected with pelvic MRI quick scan from the anticipated detection rate of 40%

SECONDARY OUTCOMES:
Detection of clinically significant prostate cancer using 3D T2 SPACE | Up to 1 year
  Number of patients with positive prostate cancer detection using 3D T2 SPACE
Detection of clinically significant prostate cancer using 3D T2 HASTE | Up to 1 year
  Number of patients with positive prostate cancer detection using 3D T2 HASTE

OTHER OUTCOMES:
Pathology specimen correlation with MRI findings | Up to 1 year
  Statistical correlation of MRI findings with final pathology specimens in those patients who elect to be treated with radical prostatectomy for treatment of their biopsy detected prostate cancer with 0 showing no correlation and 1 showing perfect correlation between findings.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Abouassaly, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- University Hospitals, Case Comprehensive Cancer Center, Cleveland, Ohio, United States